CLINICAL TRIAL: NCT06417424
Title: A Prospective, Randomized, Double-blind Controlled Clinical Study of Observation the Effect of Gastrointestinal External Stimulation on Intestinal Tract Cleaness in Patients With Senile Constipation
Brief Title: Observe Intestinal Tract Cleaness of Senile Constipation Patients Used Gastrointestinal External Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DFSC-2023(CR)-077
Record Dates: First submitted 2024-01-30; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Electric Stimulation
Keywords: ntestine cleanliness; senile constipation patients; Gastrointestinal External Stimula

STUDY DESIGN:
Intervention Model Description: 1. Received both gastrointestinal external stimulation and transcutaneouselectrical acupoint stimulation; 2. Received gastrointestinal external stimulation singly; 3. Received transcutaneouselectrical acupoint stimulation singly; 4. No stimulation was given. All groups received oral administration of polyethylene glycol for intestinal cleansing.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The Participants, investigators and outcomes Assessor don't know receiverd which intervention, only care Providers know it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- experimental group 1 (Experimental): Received both gastrointestinal external stimulation and transcutaneouselectrical acupoint stimulation for 3 days, and then oral administration of polyethylene glycol for intestinal cleansing.
  Interventions: Device: gastrointestinal external stimulation
- experimental group 2 (Experimental): Received gastrointestinal external stimulation singly, and then oral administration of polyethylene glycol for intestinal cleansing.
  Interventions: Device: gastrointestinal external stimulation
- experimental group 3 (Experimental): Received transcutaneouselectrical acupoint stimulation singly, and then oral administration of polyethylene glycol for intestinal cleansing.
  Interventions: Device: gastrointestinal external stimulation
- Control (No Intervention): No stimulation was given. Oral administration of polyethylene glycol for intestinal cleansing.

INTERVENTIONS:
Device: gastrointestinal external stimulation — We used the device Gastrointestinal multifunctional therapeutic instrument. The positive pole was placed 1 to 2cm above the umbilicus, and the negative pole was placed 4 to 10 cm to the right of the midpoint between the xiphoid process and the umbilicus.
  Arms: experimental group 1; experimental group 2; experimental group 3

SUMMARY:
This is a prospective, randomized, double-blind controlled trial. Elderly patients with constipation requiring colonoscopy were randomly divided into four groups: 1. Received both gastrointestinal external stimulation and transcutaneouselectrical acupoint stimulation; 2. Received gastrointestinal external stimulation singly; 3. Received transcutaneouselectrical acupoint stimulation singly; 4. No stimulation was given. All groups received oral administration of polyethylene glycol for intestinal cleansing. Boston Bowel Preparation Scale (BBPS) score was used to assess the quality of intestinal cleanliness , with a total score of 9, and higher scores indicating better intestinal cleanliness, and BBPS≥6 was defined effective.

DETAILED DESCRIPTION:
The early detection of intestinal lesions is extremely important, and the quality of intestine cleanliness is an important factor for the quality of colonoscopy. The elderly are at high risk of intestinal diseases. However, surveys have found that the overall quality of bowel cleanliness in elderly patients undergoing colonoscopy is poor, which affects the detection rate of colon lesions. This is a prospective, randomized, double-blind, controlled clinical trial to observe whether combined gastrointestinal surface stimulation and transcutaneous electrical acupoint stimulation can improve the quality of bowel cleansing and increase the detection rate of intestinal diseases. Elderly patients with constipation requiring colonoscopy were randomly divided into four groups: 1. Received both gastrointestinal external stimulation and transcutaneouselectrical acupoint stimulation; 2. Received gastrointestinal external stimulation singly; 3. Received transcutaneouselectrical acupoint stimulation singly; 4. No stimulation was given. All groups received oral administration of polyethylene glycol for intestinal cleansing. Boston Bowel Preparation Scale (BBPS) score was used to assess the quality of intestinal cleanliness , with a total score of 9, and higher scores indicating better intestinal cleanliness, and BBPS≥6 was defined effective.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60-80 years old;
2. Colonoscopy was planned;
3. The diagnosis of constipation was in accordance with Rome Ⅳ criteria.

Exclusion Criteria:

1. Acute myocardial infarction (within 6 months), severe heart failure (New York Heart Association class II-V, chronic renal failure (CKD stage II-V), or mental disorder;
2. Colorectal resection;
3. Drugs of aspirin, warfarin, or other anticoagulants, and coagulopathy;
4. Oral administration any drugs that may affect gastrointestinal motility, such as proton pump inhibitors, non-steroidal anti-inflammatory drugs or antibiotics (within 4 weeks), probiotics (within 2 weeks);
5. The following diseases：inflammatory bowel disease, frequent diarrhea, severe gastroparesis, intestinal perforation or obstruction;
6. Participating in other clinical trials.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale (BBPS) | 1 year
  Boston Bowel Preparation Scale (BBPS) score was used to assess the quality of intestinal cleanliness , with a total score of 9, and higher scores indicating better intestinal cleanliness, and BBPS≥6 was defined effective.
The positive rate of intestinal diseases | 1 year
  The positive rate of intestinal diseases including polyps, adenoma, adenocarcinoma, enteritis, inflammatory bowel disease,diverticulum and so on by electronic colonoscopy.

SECONDARY OUTCOMES:
Adverse reactions | 1 year
  The adverse reactions included abdominal distension, pain, nausea, vomiting, and fatigue.
Willingness to repeat | 1 year
  The Likert scale was used to judge willingness to repeat the same interventions of intestinal cleansing in future electronic colonoscopies.
Gut microbiome alterations | 1 year
  Collected fresh fecal samples before and 3 days after electrical stimulation, high-throughput sequencing was used to detect intestinal microbiome , analyzed the changes .
Gastrointestinal hormone | 1 year
  The serum levels of gastrointestinal hormones including substance P, motilin，ghrelin，growth hormone, neurotensin and vasoactive intestinal peptide were measured before and after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai easthospital, Shanghai, Pudong New Area, China

IPD SHARING:
Plan to Share IPD: Yes